CLINICAL TRIAL: NCT06541470
Title: IMAGE-GUIDED PLEURAL NEEDLE BIOPSY IN THE DIAGNOSIS OF PLEURAL DISEASES: ABRAMS NEEDLE OR CUTTING NEEDLE
Brief Title: Image-Guided Pleural Needle Biopsy in Pleural Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Muzaffer Metintas, Prof. MD, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 03.03.2022.01
Record Dates: First submitted 2024-07-10; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Biopsy; Diagnosis; Pleura; Exudate
Keywords: Pleura,; Biopsy; Ultrasonography
MeSH Terms: conditions — Disease

STUDY DESIGN:
Intervention Model Description: Prospective randomized, parallel controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Cutting needle biopsy (Other): Patients with pleural disease underwent US-assisted cutting needle biopsy.
  Interventions: Procedure: Cutting needle biopsy
- Arm B: Abrams needle biopsy (Other): Patients with pleural disease underwent US-assisted Abrams needle biopsy.
  Interventions: Procedure: Abrams needle biopsy

INTERVENTIONS:
Procedure: Cutting needle biopsy — Effectivity, reliability and safety of pleural needle biopsy in histopathological diagnosis of pleural diseases.
  Arms: Arm A: Cutting needle biopsy
Procedure: Abrams needle biopsy — Effectivity, reliability and safety of pleural needle biopsy in histopathological diagnosis of pleural diseases.
  Arms: Arm B: Abrams needle biopsy

SUMMARY:
In recent observational studies show that ultrasound guidance generally increases the success of pleural needle biopsies, it has been shown that the diagnostic success of needle biopsies is compromised and increased when the presence of pleural fluid is associated with a pleural lesion or pleural thickening or pleural nodular lesions. There is no evidence to support a common view on which needle is appropriate in which situation in terms of diagnostic success, reliability of benign diagnoses, and safety of side effects. This study aimed to compare and evaluate the diagnostic yield of the Abrams biopsy needle and the cutting biopsy needle in US-guided pleural needle biopsy to determine which needle is appropriate in which situation. As a result of the study, the diagnostic yield of the cutting needle was found to be higher in cases with pleural thickening of 1 cm or more, and the diagnostic yield of the Abrams needle was found to be higher in patients with pleural thickening of less than 1 cm.

DETAILED DESCRIPTION:
AIM A significant proportion of the most common exudative pleural effusions, approximately 40-50%, remain undiagnosed despite repeated thoracentesis and associated diagnostic procedures, including cytology. Histopathological analysis is often required for definitive diagnosis in these patients. For histopathological examination, medical thoracoscopy is generally considered to be the most effective and reliable method of obtaining tissue. However, many studies have shown that image-guided/assisted pleural needle biopsies also have a high diagnostic yield.

In recent years, respiratory physician-guided thoracic ultrasound (TUS) has become increasingly popular due to its contribution to managing pleural disease. TUS successfully guide pleural needle biopsies. Although the observational studies show that ultrasound guidance generally increases the success of needle biopsies, it has been shown that the diagnostic success of needle biopsies is compromised and increased when the presence of pleural fluid is associated with a pleural lesion or pleural thickening or pleural nodular lesions. There is no evidence to support a common view on which needle is appropriate in which situation in terms of diagnostic success, reliability of benign diagnoses, and safety of side effects. This study aimed to compare and evaluate the diagnostic yield of the Abrams biopsy needle and the cutting biopsy needle in US-guided pleural needle biopsy to determine which needle is appropriate in which situation.

METHODS This study was a prospective, randomized, parallel-group study. The Consolidated Standards of Reporting Trials (CONSORT) guidelines were followed for the study protocol. The study was conducted in the Department of Chest Diseases, Faculty of Medicine, Eskisehir Osmangazi University, and Lung and Pleural Cancer Research and Clinical Center from June 2022 to June 2023. The study was approved by the Ethical Committee of Eskisehir Osmangazi University (03.03. 2022/01) and the Ministry of Health ((E-66175679-514.04.01-800014) and was conducted according to the principles of the Declaration of Helsinki. Patients were thoroughly informed before randomization, and their written consent was obtained.

The study included one hundred and seventy-four patients who met the inclusion criteria. Before randomization, all patients underwent contrast-enhanced omputed tomography (CT).

The patients were divided into two groups: The cutting needle group (group A) and the Abrams needle group (group B). Randomization was performed on the subjects enrolled in the study. Block randomization was used with a sequence of 6.

Needle biopsies were performed in the pulmonary endoscopy suite. The biopsy was performed on the endoscopy table. Biopsy was performed using the freehand technique under US guidence. First, the pleural lesion/thickening area the needle could reach was determined as the entry point with the convex probe. The needle entry site was marked on the patient's chest wall immediately before the biopsy. The entry site was then assessed for the safety of the procedure concerning injury to major blood vessels and viscera using the US technique. Tissue sampling was performed according to standard cutting and Abrams needle procedures. After the biopsy procedures, pneumothorax was checked by the US, bleeding complications were checked by Doppler US, and control thoracentesis was performed if necessary.

Patients whose histopathological analyses after needle biopsy did not provide a specific diagnosis and whose diagnosis was reported as fibrinous pleuritis (non-specific pleuritis) were referred for medical or video thoracoscopy, depending on their preference. Patients who has fibrinous pleuritis were followed for at least 12 months. Patients with recurrent symptoms and clinical or radiological signs of disease were re-evaluated during the follow-up period, and invasive diagnostic procedures were repeated as needed. Patients who died or were lost to follow-up during this period were excluded from the analyses.

Histopathological analysis were performed by the same pathologist in the Eskisehir Osmangazi University Medical Faculty Pathology Department with histologic and immonohistochemical investigations.

Statistical analysis:

Study data were recorded in a purpose-designed case report form. A specific database was created, and SPSS version 15.0 (SPSS Inc. Chicago, Illinois) was used for statistical analysis. Patient characteristics were reported as means and percentages using descriptive statistics. The t-test, χ2 test, and two-sided Fisher's exact test were used to compare the groups. The primary endpoint of this study was the determination of sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), negative likelihood ratio (LR), and accuracy values with their confidence intervals (CIs) and complication rates of both methods concerning the diagnosis of pleural disease. These values were determined using MedCalc statistical software (version 19.1.16, MedCalc Software Software Ltd, Ostend, Belgium). In the post hoc power analysis, the power of the study was calculated as 95%. ITT (intention-to-treat) analysis was performed to show the effect of dropouts in the randomized groups.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of exudative pleural effusion for which a specific diagnosis could not be established by clinical, radiological, laboratory, and cytological examination
* Patients who do not have a high risk of side effects or contraindications for the procedures in question (without bleeding diathesis, who can be positioned appropriately for the biopsy procedure)
* Willingness to participate in the study
* Willingness to undergo an invasive procedure
* Willingness to undergo written consent for randomization and participation in the study.

Exclusion Criteria:

* Presence of parapneumonic effusion
* Patients with consciousness problems
* Any contraindication to pleural biopsy (patients with pathology in the chest wall biopsy site (infection) that would preclude biopsy, patients who are taking blood thinners (anticoagulants/antiaggregants) and cannot be interrupted for the procedure to be performed or can be interrupted by bridging with another blood thinner.)
* Any other systemic disease that could interfere with thoracic computed tomography or ultrasonography assessment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2024-02-11 (Actual); Study Completion 2024-06-02 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield of pleural needle biopsy | 12 months
  Diagnostic accuracy, sensitiviy and -LR of pleural needle biopsies with cutting or Abrams needle biopsy.

SECONDARY OUTCOMES:
Safety of pleural needle biopsy | 12 months
  Determining of the complications for pleural needle biopsies with cutting or Abrams needle biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Emre Celik, MD, Principal Investigator — Eskisehir Osmangazi University Medical Faculty
Locations (5):
- Turkey (Türkiye) (5):
  - ESOGU Medical Faculty Department of Chest Diseases, Eskişehir, Meselik - Eskisehir
  - Muzaffer Metintas, Eskişehir, Meselik
  - Selma Metintas, Eskişehir, Meselik
  - ESOGU Lung and Pleural Cancers Clinical and Research Center, Eskişehir, Meselik
  - Eskisehir Osmangazi University Medical Faculty Department of Chest Diseases, Eskişehir, Tepebaşı

IPD SHARING:
Plan to Share IPD: Yes
INFORMATION ABOUT THE STUDY SUCH AS METHOD, CASES AND RESULTS WILL BE SENT IF REQUESTED.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2 MONTHS AFTER PUBLICATION
Access Criteria: Optional
URL: http://ogu.edu.tr